CLINICAL TRIAL: NCT00875264
Title: An Open-Label Study to Determine the Maximum Tolerated Oral Dose of the Kinase Inhibitor CEP-11981 in Patients With Advanced Cancer
Brief Title: Open-Label Study to Determine the Maximum Tolerated Oral Dose of the Kinase Inhibitor CEP-11981 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C11981/1047/ON/US
Record Dates: First submitted 2009-04-01; First posted 2009-04-03 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Cancer
Keywords: CEP-11981; TIE-2; VEGF-R
MeSH Terms: conditions — Neoplasms | interventions — 11-(2-methylpropyl)-12,13-dihydro-2-methyl-8-(pyrimidin-2-ylamino)-4H-indazolo(5,4-a)pyrrolo(3,4-c)carbazol-4-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): At least one 6-week (42-day) cycle in which patients will be treated daily with CEP-11981 for 28 days, followed by a treatment-free period of 14 days.
  Interventions: Drug: CEP-11981 (kinase inhibitor)

INTERVENTIONS:
Drug: CEP-11981 (kinase inhibitor) — Patients will be treated with oral CEP-11981 once daily for 28 days, followed by a treatment-free period of 14 days. This 42-day (6-week) period will constitute 1 cycle. The starting dose for the study will be 3 mg/m2. Dose escalation from this starting dose follows a modified Fibonacci sequence.

SUMMARY:
The primary objective of this study is to determine the maximum tolerated dose (MTD) and dose-limiting toxicities of CEP-11981 in patients with advanced, relapsed/refractory solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

The patient:

* has a histologically or cytologically confirmed solid tumor that has relapsed or is refractory. Additionally, the tumor must be considered unresponsive or poorly responsive to accepted treatment modalities.
* has a life expectancy of at least 12 weeks.
* has an Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1, or 2.
* has normal neurologic examination findings. Patients having neurologic signs and symptoms indicative of brain metastases must undergo magnetic resonance imaging (MRI) to rule out brain metastases.
* has fully recovered from any prior surgical procedure(s).
* has fully recovered from reversible side effects of prior therapy for cancer including radiation therapy, chemotherapy, and immunotherapy.
* is in appropriate health as determined by medical and psychiatric history, medical examination, electrocardiography (ECG), serum chemistry and hematology tests, and urinalysis.
* if a woman of childbearing potential (not surgically sterile or who are not 2 years postmenopausal), must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study. Acceptable methods of contraception include abstinence, barrier method with spermicide, intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method.
* if a man, not surgically sterile or who is capable of producing offspring, must practice abstinence or use a barrier method of birth control, and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study.
* is willing and able to comply with study restrictions and to return to the clinic for evaluations (including follow-up).

Key Exclusion Criteria:

The patient:

* has any of the following hematologic values: absolute neutrophil count (ANC) less than 1500/mm3, platelet count less than 100000/mm3, hemoglobin less than 9 g/dL.
* has any of the following hepatic function values: bilirubin greater than 1.5 times the upper limit of normal (ULN), alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2.0 times the ULN in the absence of known hepatic metastases, or ALT or AST greater than 3.0 times the ULN in the presence of known hepatic metastases.
* has a serum creatinine value greater than 1.5 mg/dL.
* has known cerebral metastases.
* is currently on warfarin or heparin therapy.
* has any pre-existing coagulopathy, recent hemoptysis, gross hematuria, or gastrointestinal bleeding, and a history of a clinically significant cardiovascular or cerebrovascular event within 6 months prior to study entry.
* has uncontrolled hypertension defined as a blood pressure measurement greater than 150 mm Hg systolic or 90 mm Hg diastolic with medication.
* is receiving any other antineoplastic treatment for solid tumors. (Continuing hormonal treatment is permitted.)
* has received any investigational drug within the past 4 weeks.
* has previously been enrolled in the study or received CEP-11981.
* has known hypersensitivity to gelatin or lactose monohydrate.
* is a woman who is pregnant or lactating.
* has taken a medication known to be a potent inducer of CYP1A2, CYP2C8, or CYP3A4 within 4 weeks prior to the first dose of study drug.
* has taken a medication known to be a potent inhibitor of CYP1A2, CYP2C8, or CYP3A4 within 2 weeks prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs) of CEP-11981, as defined in the Study Protocol. | At least one 6-week (42-day) cycle, which includes 28 days treatment during each cycle

SECONDARY OUTCOMES:
Tumor response or progression using Response Evaluation Criteria in Solid Tumors (RECIST) criteria. | At least one 6-week (42-day) cycle, which includes 28 days treatment during each cycle
Measurement of Pharmacokinetic parameters | Cycle 1 (42 days) and Day 1 of Cycle 2
Safety and tolerability of CEP-11981 | At least one 6-week (42-day) cycle, which includes 28 days treatment during each cycle

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon